CLINICAL TRIAL: NCT03357419
Title: A Randomized, Placebo Controlled Trial of the Effect of Prophylactic Antibiotics on Surgical Site Infection Lower Limb Skin Excisions
Brief Title: The Effect of Prophylactic Antibiotics on Surgical Site Infection Lower Limb Skin Excisions
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulties in production placebo antibiotics
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0569-17 RMB
Record Dates: First submitted 2017-11-23; First posted 2017-11-29 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Skin Lesion
MeSH Terms: interventions — Cephalexin; Clindamycin

STUDY DESIGN:
Intervention Model Description: A randomized, 1:1, double-blind, placebo controlled trial designed to evaluate the effect of prophylactic antibiotic on patients presenting for skin excision from lower limbs.
  Before the surgery patient's demographics, medical history, skin lesion's site, properties and size will be documented. During the surgery the size of the wound and the sutures used will be documented. Afterwards, the wound will be assed for signs of infection (criteria adapted from the Centre for Disease Control and Prevention definition for superficial SSI [42]) and other complications during the follow-up period as needed until sutures will be removed at our clinic.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prophylactic antibiotic (Active Comparator): Each active arm patient will be given the tested drug on admission, 30-60 minutes before the surgery, by the nurses.
  2 g dose of cephalexin (or Clindamycin 600 mg for patients suffering from allergy) will be given once, orally, 30-60 minutes prior to skin lesion excision
  Interventions: Drug: Cephalexin
- placebo oral capsule (Placebo Comparator): Each placebo arm patient will be given the placebo drug on admission, 30-60 minutes before the surgery, by the nurses
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Cephalexin — The subjects will be randomized, at the operation day, to one of two treatment groups:
  * group 1: prophylactic antibiotic
  * group 2: placebo oral capsule
    * Sealed envelopes, numbered according to the randomization dose, containing the drug or placebo will be prepared in advance and provided to the patient following randomization.
    * Each patient will be given the randomized drug on admission, 30-60 minutes before the surgery, by the nurses.
  Other Names: Clindamycin hydrochloride
  Arms: prophylactic antibiotic
Drug: Placebo oral capsule — The subjects will be randomized, at the operation day, to one of two treatment groups:
  * group 1: prophylactic antibiotic
  * group 2: placebo
    * Sealed envelopes, numbered according to the randomization dose, containing the drug or placebo will be prepared in advance and provided to the patient following randomization.
    * Each patient will be given the randomized drug on admission, 30-60 minutes before the surgery, by the nurses.
  Arms: placebo oral capsule

SUMMARY:
The incidence of surgical site infection (SSI) infection in clean dermatologic surgery is very low, between 1-3%. Studies have demonstrated a much higher infection rate in skin excision surgeries in the lower limbs, up to 10% in most studies, and even 35.7% infection rate in a recent study from Australia.

To our knowledge, there are no clinical trials demonstrating the efficacy of prophylactic antibiotic given prior to skin lesion excision from the lower limbs.

DETAILED DESCRIPTION:
The majority of skin cancers are treated by surgical excision which is being performed in outpatient and primary care settings.

Surgical site infection (SSI) is one of the few complications of this relatively minor surgery. These infections often require antibiotics and repeat consultations to assess wound healing. Moreover, they can potentially lead to significant bacteremic complications and impair cosmetic outcome.

The incidence of surgical site infection (SSI), bacterial endocarditis, and joint prosthesis infection in clean dermatologic surgery is very low. This is reflected in skin lesion excisions, with a rate of between 1% and 3% in most studies.

Indiscriminate use of antibacterials is causing multidrug-resistant bacteria to emerge. Furthermore, antibacterials can cause anaphylactic reactions and even death in rare cases. There are also known interactions between several medications taken long term for underlying health problems and antibacterials.[ Therefore the routine use of antibiotics is not recommended. Despite this, medical practitioners vary greatly in their use of antibacterial prophylaxis and frequently overprescribe antibacterials for the prevention of SSI, bacterial endocarditis, and prosthesis infection.

Overall, rates of wound infection in cutaneous surgery are generally very low in clean wounds, with 1-3% quoted in most studies.

A study involving 5091 skin surgery cases with an overall infection rate of 1.47% found SSI rates >5% below the knee (6.92%), in the groin area (10%), for wedge excisions of the lip and ear (8.57%), and for grafts (8.7%).Other studies have confirmed higher infection rates below the knee,in the groin,and on the thighs, legs, and feet.

A well designed study in subtropical Australia found infection rates as high as 8.6%,which calls into question the role of humidity and ambient temperature in postoperative dermatologic infection.

Wounds can be classified (class I-IV) according to the site and status of the wound preoperatively (table I). This classification, based on the 1985 Centers for Disease Control (CDC) guidelines for prevention of surgical wound infections,has been found to be a strong predictor of subsequent infection rates.

The need for prophylactic antibacterials depends on the wound classification.Class I wounds (primary closure of wounds on clean, non-contaminated skin under sterile conditions) should generally not receive antibacterial prophylaxis.

The 1992 CDC definitions of nosocomial infections give clear guidelines for diagnosing SSI.Superficial surgical site skin infection can be diagnosed if it involves skin, subcutaneous tissues, or muscle above the fascial layer at the incision site, it occurs within 30 days of surgery, and at least one of the following is present:

* Purulent discharge from the incisional wound.
* Organisms are isolated on culture of aseptically obtained wound fluid or tissue.
* One or more of the following is present: pain, tenderness, localized swelling, redness, heat.
* The surgeon deliberately reopens the wound (unless culture of the incision is negative).
* The treating doctor diagnoses a superficial incisional SSI. Even with the use of guidelines, the definition of wound infection is subject to considerable inter- and intra-observer variation.

Staphylococcus aureus and Streptococcus pyogenes are the most common pathogens causing wound infection in keratinized skin.Other microorganisms causing SSI include coagulase-negative staphylococci, Enterococcus spp., Pseudomonas aeruginosa, and Enterobacter spp.

Evidence suggests the following to be risk factors for postoperative wound infections: poor nutritional status obesity, smoking and diabetes mellitus. Other studies have shown the excisions of skin cancers may be complicated by higher infection rate.

Surgical risk factors include Potential sources of microbial contamination of the surgical wound include the patient's skin, flora of the skin and nares of the operating team, the surgical apparel, the surgeons' gloves, and airborne organisms in the operating room.

Surgical technique is also an important, studies have shown that excessive tissue injury and high-tension closure are risk factors for SSI. Other studies have demonstrated that satisfactory control of hemostasis helps prevent SSI. Two prospective multivariate analyses, one with 3788 surgical skin procedures and the other with 3491, have shown that hemorrhagic complications in both simple and complex dermatologic surgical procedures are an independent risk factor for SSI.

Recent prospective studies categorizing wound infections according to body site and surgical technique have identified patients who may be at higher risk of infection following dermatologic surgery including surgeries below the knee, in the groin area, skin graft at any site, skin graft at any site, Wedge excision or flap surgery on the ear and lip.

However, there are no published large, randomized controlled trials measuring the effectiveness of prophylactic oral antibacterials.

One study, with an overall infection rate of 1.47%, involved 5091 surgical skin excisions in 2424 patients, none of whom received prophylactic antibacterials. Surgical procedures with an infection rate >5% were skin grafts (8.7%), and wedge excisions on the ear or lip (8.57%). Anatomic sites with a significantly higher infection rate were all areas below the knee (6.92%), and the groin (10%). A study of 857 skin procedures in tropical north Queensland, Australia, with an overall infection rate of 8.7%, found location on lower extremities to be an independent risk factor for wound infection.The infection rates in this study were 14% on the thighs and 15% on the legs and feet. Other studies have found higher infection rates below the knee and in the groin.

Prophylactic antibacterials will be most effective if present at the surgical site at the time of incision and should, therefore, be should administered prior to the procedure. Bacteria introduced during the surgical procedure reside and multiply in the wound coagulum. Since it is difficult for antibacterials to gain access to the coagulum, multiplying bacteria remain relatively protected there unless antibacterials are present prior to its formation.

Antibacterial prophylaxis, whether oral or intravenous, should be administered 30-60 minutes prior to dermatologic surgery.

There have been no large-scale, prospective trials comparing different prophylactic antibacterial regimens. Based on the organisms most likely to cause infection, the penicillinase- resistant penicillins or first-generation cephalosporins are generally the oral antibacterials of choice for SSI prophylaxis Wright et al. Recommended either cefalexin 2g or dicloxacillin 2 g administered orally 30-60 minutes before the surgical procedure for most dermatologic surgery.

Several expert groups-including the Mayo Clinic's Department of Dermatological Surgery-have suggested that a single oral dose of perioperative antibiotic prophylaxis may be indicated in certain 'high risk' situations such as excisions from the lower limb. If effective, this may be a low-cost and easily implemented method of reducing the incidence of SSI in selected situations. A small prospective randomized placebo controlled double blind trial, by Smith et al, from Australia, on patients undergoing skin excision of lesions in the lower limb, have compared the difference in infection rate between patients given prophylactic Cephalexin (n=24) having incidence of SSI of 12.5%, compared to the placebo group (n=28) with incidence of SSI of 35.7%. The reduction was not statistically significant (p=0.064).

To our knowledge, there are no clinical trials demonstrating the efficacy of prophylactic antibiotic given prior to skin lesion excision from the lower limbs.

This trial sought to determine the efficacy of a 2 g dose of cephalexin given 30-60 min prior to skin lesion excision from the lower limb in preventing the subsequent development of an SSI.

ELIGIBILITY:
Inclusion Criteria:

Patients presenting for skin excision from the thigh, shin or foot, in the Rambam medical center

Exclusion Criteria:

* Younger than 18 years old.
* Not capable of providing informed consent.
* Declined to participate.
* Currently taking antibiotics.
* Surgeon feels they are clinically indicated for antibiotic treatment following excision.
* Lesions considered as contaminated/ infected prior to surgery.
* Excision not utilizing primary closure or skin graft.
* Patient unable to return for suture removal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2022-03-27 (Actual)

PRIMARY OUTCOMES:
The primary end point is absence of infection after 1 month follow-up. | 1-2 years
  Wounds will be assessed for infection by the doctor at the time of removal of sutures, or sooner if the patient had complaints about the wound.
  The definition of SSI and its classification to superficial or deep will be based on the presence of any of the following criteria that were adapted from the Centre for Disease Control and Prevention (CDC) definition for superficial SSI [42]. The primary outcome will consist of any SSI, superficial or deep.

CONTACTS AND LOCATIONS:
Overall Officials: Yehuda Ullmann, Proffesor, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Department of Plastic Surgery, Rambam Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wright TI, Baddour LM, Berbari EF, Roenigk RK, Phillips PK, Jacobs MA, Otley CC. Antibiotic prophylaxis in dermatologic surgery: advisory statement 2008. J Am Acad Dermatol. 2008 Sep;59(3):464-73. doi: 10.1016/j.jaad.2008.04.031. PMID 18694679
- [Background] Maragh SL, Otley CC, Roenigk RK, Phillips PK; Division of Dermatologic Surgery, Mayo Clinic, Rochester, MN. Antibiotic prophylaxis in dermatologic surgery: updated guidelines. Dermatol Surg. 2005 Jan;31(1):83-91. doi: 10.1111/j.1524-4725.2005.31014. PMID 15720101
- [Background] Rogues AM, Lasheras A, Amici JM, Guillot P, Beylot C, Taieb A, Gachie JP. Infection control practices and infectious complications in dermatological surgery. J Hosp Infect. 2007 Mar;65(3):258-63. doi: 10.1016/j.jhin.2006.09.030. Epub 2007 Jan 22. PMID 17244515
- [Background] Horan TC, Gaynes RP, Martone WJ, Jarvis WR, Emori TG. CDC definitions of nosocomial surgical site infections, 1992: a modification of CDC definitions of surgical wound infections. Infect Control Hosp Epidemiol. 1992 Oct;13(10):606-8. No abstract available. PMID 1334988
- [Background] Mangram AJ, Horan TC, Pearson ML, Silver LC, Jarvis WR. Guideline for Prevention of Surgical Site Infection, 1999. Centers for Disease Control and Prevention (CDC) Hospital Infection Control Practices Advisory Committee. Am J Infect Control. 1999 Apr;27(2):97-132; quiz 133-4; discussion 96. PMID 10196487
- [Result] Dixon AJ, Dixon MP, Askew DA, Wilkinson D. Prospective study of wound infections in dermatologic surgery in the absence of prophylactic antibiotics. Dermatol Surg. 2006 Jun;32(6):819-26; discussion 826-7. doi: 10.1111/j.1524-4725.2006.32167.x. PMID 16792648
- [Result] Amici JM, Rogues AM, Lasheras A, Gachie JP, Guillot P, Beylot C, Thomas L, Taieb A. A prospective study of the incidence of complications associated with dermatological surgery. Br J Dermatol. 2005 Nov;153(5):967-71. doi: 10.1111/j.1365-2133.2005.06861.x. PMID 16225607
- [Result] Burke JP. Maximizing appropriate antibiotic prophylaxis for surgical patients: an update from LDS Hospital, Salt Lake City. Clin Infect Dis. 2001 Sep 1;33 Suppl 2:S78-83. doi: 10.1086/321861. PMID 11486303
- [Result] Smith SC, Heal CF, Buttner PG. Prevention of surgical site infection in lower limb skin lesion excisions with single dose oral antibiotic prophylaxis: a prospective randomised placebo-controlled double-blind trial. BMJ Open. 2014 Jul 30;4(7):e005270. doi: 10.1136/bmjopen-2014-005270. PMID 25079934